CLINICAL TRIAL: NCT03439436
Title: An Observer-blind, Multi-centre, Randomized, Parallel-group Study to Compare the Efficacy and Safety of Two Formulations of Xylometazoline/Dexpanthenol Nasal Spray for the Treatment of Nasal Congestion.
Brief Title: A Study to Compare Two Formulations of Xylometazoline/Dexpanthenol Nasal Spray for the Treatment of Nasal Congestion.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CO-170117145845-URCT
Record Dates: First submitted 2018-01-15; First posted 2018-02-20 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Nasal Congestion
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Bottles kept in neutral outer boxes. Staff performing assessments kept unaware of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- xylo+dex nasal spray (0.1 mg+5 mg/dose) (Experimental): Xylometazoline+Dexpanthenol metered nasal spray (0.1 mg+5 mg/dose) for nasal congestion. One spray into each nostril, 3 times daily for max 5 days.
  Interventions: Drug: xylo+dex nasal spray (0.1 mg+5 mg/dose)
- Nasic (Active Comparator): Xylometazoline+Dexpanthenol metered nasal spray (0.1 mg+5 mg/dose) for nasal congestion. One spray into each nostril, 3 times daily for max 5 days.
  Interventions: Drug: Nasic

INTERVENTIONS:
Drug: xylo+dex nasal spray (0.1 mg+5 mg/dose) — Xylometazoline+Dexpanthenol metered nasal spray (0.1 mg+5 mg/dose) for nasal congestion. One spray into each nostril, 3 times daily for max 5 days.
  Other Names: xylo+dex metered nasal spray (0.1 mg+5 mg/dose)
  Arms: xylo+dex nasal spray (0.1 mg+5 mg/dose)
Drug: Nasic — Xylometazoline+Dexpanthenol metered nasal spray (0.1 mg+5 mg/dose) for nasal congestion. One spray into each nostril, 3 times daily for max 5 days.
  Other Names: xylo+dex metered nasal spray (0.1 mg+5 mg/dose)
  Arms: Nasic

SUMMARY:
An observer-blind, multi-centre, randomized, parallel-group study to compare the efficacy and safety of two formulations of xylometazoline/dexpanthenol nasal spray for the treatment of nasal congestion caused by an acute upper respiratory tract infection in adults.

DETAILED DESCRIPTION:
This observer-blind multi-center, randomized, parallel-group study in adults is designed to demonstrate non-inferiority between two formulations of xylometazoline/dexpanthenol nasal sprays in terms of efficacy and safety, when the products are used according to labeled instructions in a home based setting.

Subjects suffering from nasal congestion caused by acute Upper Respiratory Tract Infection (URTI) and seeking medical counselling, will after screening and baseline assessment of nasal congestion, be randomized, and perform additional baseline subjective assessments of nasal rhinorrhea (scores on categorical scales). The Investigator will perform subjective baseline assessments of crust formation and dryness, redness and edema of nasal mucosa (anterior rhinoscopy using nasal speculum or otoscope).

After the baseline assessments, the subjects will receive xylometazoline/dexpanthenol nasal spray or marketed reference nasal spray according to randomization.The first dose will be taken at the site under supervision. The study nurse will schedule visits for 24 hours, 72 hours and 120 hours after this first dose and the subjects will be released for home based treatment. At the 72-hour visit, the primary and secondary efficacy endpoints will be assessed by the subject and the Investigator, safety will be followed up and subjects will also evaluate the treatment in a global assessment. At the 24-hour visit and at the final visit, after a maximum of 5 full days (120 hours) of treatment, all secondary endpoints will be assessed and safety will be followed up.

ELIGIBILITY:
Inclusion Criteria

* Subjects of 18 years of age or older;
* Subjects suffering from nasal congestion with a clinical diagnosis of acute upper respiratory tract infection where symptoms of nasal congestion have persisted for minimum of 3 hours and maximum of 36 hours;
* Body mass index (BMI) 18.5 to 35 (inclusive) at screening;
* Indicate at least moderate congestion on a categorical scale ranging from (0) none, (1) mild, (2) moderate, (3) severe or (4) very severe, completed at screening and at baseline;
* Females of childbearing potential must have a negative urine pregnancy test at screening;
* Male and non-pregnant, non-lactating females must agree to the contraceptive requirements (including female partners' use of highly effective form of birth control for at least 3 months before the study, during the study and up to 30 days after the last dose of investigational products) as outlined in protocol.
* Are able and willing to comprehend and follow the requirements of the study (including availability on scheduled visit dates) based upon research site personnel´s assessment;
* Are able to read and understand the local language;
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study and consents to participate.

Exclusion Criteria

* Females who are pregnant, breastfeeding or trying to conceive;
* Male with a pregnant partner or a partner who is currently trying to conceive;
* Have a known allergy or hypersensitivity to xylometazoline, dexpanthenol or any of the excipients of the formulations;
* Presence or history of a medical condition in the investigator's opinion that may jeopardize the subject´s safety or well-being, or the integrity of the study (e.g., hepatic, renal, pancreatic, gastrointestinal, cardiovascular, cerebrovascular, thyroid, seizure, asthma, allergy, drug intolerance, or psychiatric disorders; uncontrolled hypertension indicated as systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg; or uncontrolled diabetes in the last 6 months);
* Suspected alcohol or substance abuse (e.g., amphetamines, benzodiazepines, cocaine, marijuana, opiates);
* Clinically significant laboratory abnormality that cannot be explained by the acute upper respiratory tract infection;
* Presenting axillary temperature of 38.5 Celsius degrees or above;
* Acute and/or chronic respiratory tract disease or other concomitant disease with potential to compromise breathing (asthma, bronchopneumonia);
* Chronic ear, nose and throat (ENT) conditions e.g. nasal polyps, perennial or seasonal allergic rhinitis, or significant nasal septum deviation;
* Suspected fungal upper respiratory tract infection e.g., candida infection;
* Known or suspected bacterial upper respiratory tract infection or purulent pharyngitis;
* Have contraindicated conditions: arterial hypertension, tachycardia, marked atherosclerosis, atrophic rhinitis, rhinitis sicca, hyperthyroidism, porphyria, prostatic hyperplasia, glaucoma, previous surgical intervention on the meninges;
* Are currently taking monoamine oxidase inhibitors (MAOIs) or tricyclic antidepressants;
* Use of any analgesic, antipyretic or "cold and flu" medication including non-prescription medication and/or herbal products within previous 8 hours, for naproxen containing products within previous 12 hours;
* Use of any nasal or oral decongestant including non-prescription medication and/or herbal products for the presenting episode of nasal congestion;
* Use of any menthol containing medications or confectionary including non-prescription medication and/or herbal products within 6 hours of baseline;
* Participation in any interventional clinical trials within 30 days before screening or had previous participation in this trial;
* Subjects who are related to those persons involved directly or indirectly with the conduct of this study (i.e., Principal Investigator, sub-investigators, study coordinators, other site personnel, employees of Johnson & Johnson subsidiaries, contractors of Johnson & Johnson, and the families of each).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in self-assessment of nasal congestion after 72 hours of treatment. | After 72 hours of treatment.
  Change from baseline in self-assessment of nasal congestion after 72 hours of treatment.

SECONDARY OUTCOMES:
Change from baseline in self-assessment of nasal congestion at 24 and 120 hours post dose. | At 24 and 120 hours post dose.
  Change from baseline in self-assessment of nasal congestion at 24 and 120 hours post dose.
Change from baseline in self-assessment of rhinorrhea after 24 hours, 72 and 120 hours post dose. | At 24 hours, 72 and 120 hours post dose
  Change from baseline in self-assessment of rhinorrhea after 24 hours, 72 and 120 hours post dose.
Assessment of nasal crusting after 24 hours, 72 hours and 120 hours post dose. | At 24 hours, 72 hours and 120 hours post dose.
  Assessment of nasal crusting after 24 hours, 72 hours and 120 hours post dose.
Assessment of dryness of nasal mucosa after 24 hours, 72 hours and 120 hours post dose. | At 24 hours, 72 hours and 120 hours post dose.
  Assessment of dryness of nasal mucosa after 24 hours, 72 hours and 120 hours post dose.
Assessment of redness of nasal mucosa after 24 hours, 72 hours and 120 hours post dose. | At 24 hours, 72 hours and 120 hours post dose.
  Assessment of redness of nasal mucosa after 24 hours, 72 hours and 120 hours post dose.
Assessment of edema of nasal mucosa after 24 hours, 72 hours and 120 hours post dose. | At 24 hours, 72 hours and 120 hours post dose
  Assessment of edema of nasal mucosa after 24 hours, 72 hours and 120 hours post dose.
Global evaluation assessments of study treatment by subjects at 72 hours post dose. | At 72 hours post dose.
  Global evaluation assessments of study treatment by subjects at 72 hours post dose.
Frequency and severity of treatment emergent AEs reported during the study. | Through study completion, an average of 5 months.
  Each treatment emergent AE reported during the trial and it´s severity will be tabulated in a list, capturing frequency and severity of all treatment emergent AEs occuring during the trial.
Frequency and severity of AEs possibly, probably, or very likely related to the study drug during study treatment. | Through study completion, an average of 5 months.
  Each AE which has been ranked as possibly, probably, or very likely related to the study drug during study treatment will be tabulated in a list capturing frequency and severity of all these AEs occuring during the trial.
Occurrence of serious AEs (SAEs). | Through study completion, an average of 5 months.
  Occurrence of serious AEs (SAEs), will be tabulated in a list.
Occurence of AEs resulting in pre-mature withdrawal from the study. | Througout study completion, an average of 5 months.
  Occurence of AEs resulting in pre-mature withdrawal from the study will be tabulated in a list.

OTHER OUTCOMES:
Subject compliance with the study medication dosing regimen by reporting of doses taken in subject diary. | Through study completion, an average of 5 months.
  Subject compliance with the study medication dosing regimen by reporting of doses taken in subject diary.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Lioznov, MD, Principal Investigator — The First St. Petersburg state medical University n.a. Acad. I. P. Pavlov; Tatiana E Morozova, MD, Principal Investigator — First Moscow State Medical University n. a. I. M. Sechenov; Vladimir Popov, MD, Principal Investigator — Railways clinical hospital n.a.Semashko at Lublino station JSC "RZD"; Zhanna M Sizova, MD, Principal Investigator — City Polyclinic #2; Konstantin A Zakharov, MD, Principal Investigator — "Scientific and Research centre Eco-safety" Limited Liability Company; Alison Hughes, Study Director — R&D MedClin EMEA, J&J
Locations (5):
- Russia (5):
  - Railways clinical hospital n.a.Semashko at Lublino station JSC "RZD", Moscow
  - City Polyclinic #2, Moscow
  - First Moscow State Medical University n. a. I. M. Sechenov, Moscow
  - "Scientific and Research centre Eco-safety" Limited Liability Company, Saint Petersburg
  - The First St. Petersburg state medical University n.a. Acad. I. P. Pavlov, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CO-170117145845-URCT&attachmentIdentifier=7eb88242-3fe6-41e3-83c8-ad759268502b&fileName=CO-170117145845-URCT_Full_CSR_Synopsis_.pdf&versionIdentifier=